CLINICAL TRIAL: NCT02013388
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Multiple-Ascending Dose Study Evaluating the Safety, Tolerability, and Pharmacokinetic Effects of N91115 in Healthy Subjects
Brief Title: MAD Study Evaluating the Safety, Tolerability, and Pharmacokinetic Effects of N91115 in Healthy Subjects
Acronym: SNO2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nivalis Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N91115-1H-01
Record Dates: First submitted 2013-12-09; First posted 2013-12-17 (Estimated); Results first posted 2015-03-18 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-11

CONDITIONS: Healthy
Keywords: N91115; GSNORi; SNO; Cavosonstat
MeSH Terms: interventions — cavosonstat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- 10 mg (Experimental): single oral daily dose of 10 mg N91115 for 14 days
  Interventions: Drug: N91115
- Placebo (Placebo Comparator): single oral daily dose of placebo for 14 days
  Interventions: Drug: Placebo
- 50 mg (Experimental): single oral daily dose of 50 mg N91115 for 14 days
  Interventions: Drug: N91115
- 50 mg (single dose) (Experimental): single oral dose of 50 mg N91115
  Interventions: Drug: N91115
- 250 mg (Experimental): single oral daily dose of 250 mg N91115 for 14 days (fasted)
  Interventions: Drug: N91115
- 250 mg (Fed) (Experimental): single oral daily dose of 250 mg N91115 for 1 day (fed fat meal)
  Interventions: Drug: N91115
- 500 mg (Experimental): single oral daily dose of 500 mg N91115 for 14 days
  Interventions: Drug: N91115
- Placebo-Day 1 only (Placebo Comparator): Single oral dose of placebo (Day 1 only)
  Interventions: Drug: Placebo-Day 1 only

INTERVENTIONS:
Drug: N91115 — Given PO daily for 14 days
  Other Names: Cavosonstat
  Arms: 10 mg; 250 mg; 50 mg; 500 mg
Drug: Placebo — Given PO daily for 14 days
  Arms: Placebo
Drug: N91115 — Given PO only on Day 1
  Other Names: Cavosonstat
  Arms: 250 mg (Fed); 50 mg (single dose)
Drug: Placebo-Day 1 only — Given PO- only on Day 1 (single dosed to match single dose treatments)
  Other Names: Placebo
  Arms: Placebo-Day 1 only

SUMMARY:
A study in healthy subjects to assess the safety, tolerability, and pharmacokinetics of N91115.

DETAILED DESCRIPTION:
This Phase 1 study in healthy subjects is being conducted to assess the safety, tolerability, and pharmacokinetics of N91115. Also, a comparison of the fasted versus fed with a high fat meal were compared for PK.

ELIGIBILITY:
Inclusion Criteria:

* Subject voluntarily agrees to participate in this study and signs an Institutional Review Board (IRB)-approved informed consent prior to performing any of the screening procedures and in the opinion of the PI complies with all the requirements of the study.
* Subject is healthy, determined at the screening medical evaluation (including but not limited to medical history, physical examination and clinical laboratory evaluations).
* Subject is Caucasian.
* Female subject must be of non-childbearing potential (surgically sterile [hysterectomy or bilateral tubal ligation] or post-menopausal ≥ 1 year with follicle stimulating hormone [FSH] > 40 U/L). Women receiving hormone replacement therapy (HRT) are eligible to enroll.
* Male subject must agree to use condoms and refrain from sperm donation from Day 1 until 30 days post last dose or have documentation of vasectomy.
* Subject has a body weight > 50 kg and body mass index (BMI) between 19.5 and 32 kg/m2, inclusive, at screening.
* Subject has no clinically significant abnormal findings related to their systolic or diastolic blood pressure (BP), per the investigator's judgment, at screening or Day 1.
* Subject has no clinically significant abnormal findings in 12 lead ECG, per the investigator's judgment, at screening.

Exclusion Criteria:

* Subject has clinically significant history or evidence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, immunological, or psychiatric disorder(s) as determined by the investigator or designee.
* Subject has clinically significant abnormalities on a 12 lead ECG done at screening
* Subject has clinically significant abnormalities on a 48-hour ambulatory ECG done at screening
* Subject has any disorder that would interfere with the absorption, distribution, metabolism, or excretion of drugs.
* Subject has any concurrent disease or condition that, in the opinion of the investigator, would make the subject unsuitable for participation in the clinical study.
* Subject is unlikely to comply with the protocol requirements, instructions, and study related restrictions; e.g., uncooperative attitude, unavailable for follow-up call, and/or improbability of completing the clinical study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Galloway, MD, Principal Investigator — Davita Clinical Research; Steven A Shoemaker, MD, Study Director — Nivalis Therapeutics, Inc.
Locations (1):
- DaVita Clinical Research, Lakewood, Colorado, United States

REFERENCES:
- [Derived] Donaldson SH, Solomon GM, Zeitlin PL, Flume PA, Casey A, McCoy K, Zemanick ET, Mandagere A, Troha JM, Shoemaker SA, Chmiel JF, Taylor-Cousar JL. Pharmacokinetics and safety of cavosonstat (N91115) in healthy and cystic fibrosis adults homozygous for F508DEL-CFTR. J Cyst Fibros. 2017 May;16(3):371-379. doi: 10.1016/j.jcf.2017.01.009. Epub 2017 Feb 13. PMID 28209466
- See also: Home Page — http://n30pharma.com
- See also: Phase 1 Unit — http://davitaclinicalresearch.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo-single Dose: Placebo: Given PO daily for 1 day
Period: Overall Study
Arm/Group | Placebo | 10 mg | 50 mg | 250 mg | 500 mg | 50 mg (Single Dose) | 250 mg (Fed) | Placebo-single Dose
Started | 9 | 6 | 6 | 6 | 6 | 6 | 6 | 4
Completed | 8 | 6 | 6 | 6 | 5 | 6 | 6 | 4
Not Completed | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — work emergency | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo- Single Dose: single oral dose Placebo: Given PO daily for 1day
- Total: Total of all reporting groups
Arm/Group | Placebo | 10 mg | 50 mg | 250 mg | 500 mg | 50 mg (Single Dose) | 250 mg (Fed) | Placebo- Single Dose | Total
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 6 | 6 | 6 | 4 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (12.32) | 41.3 (14.90) | 40.2 (14.25) | 39.7 (10.03) | 37.3 (10.91) | 42.3 (9.40) | 37.8 (11.84) | 41.3 (11.59) | 39.1 (11.40)
Gender [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 2 | 5 | 0 | 2 | 2 | 16
  Male | 8 | 4 | 4 | 4 | 1 | 6 | 4 | 2 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 4 | 48
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 4 | 48
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of N91115
Description: Assessments are based on numbers of subjects with abnormal clinical evaluations, abnormal laboratory assessments, and adverse events.
Time Frame: 21 Days
Population: All patients enrolled in the study were evaluated for safety endpoints
Measure: Number; unit: participants
Arm/Group | Placebo | 10 mg | 50 mg | 250 mg | 500 mg | 50 mg (Single Dose) | 250 mg (Fed) | Placebo- Single Dose
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 6 | 6 | 6 | 4
participants
  Subjects with at least one TEAE | 9 | 6 | 6 | 6 | 6 | 1 | 4 | 2
  Subjects with at least one study treatment TEAE | 5 | 4 | 4 | 2 | 2 | 1 | 0 | 1

2. Primary Outcome: Pharmacokinetics: Day 1 AUClast
Description: Day 1 AUClast plasma values from treatment groups completing 14 days of N91115 administration
Time Frame: Day 1
Population: All patients that had plasma samples collected were included in the analysis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 10 mg | 50 mg | 250 mg | 500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5
h*ng/mL | 327 (24.0) | 1530 (23.5) | 12000 (20.6) | 32400 (44.4)

3. Primary Outcome: Pharmacokinetics: AUCtau Day 14
Description: Plasma analysis of AUCtau values from the end of the dosing period (Day 14) with N91115
Time Frame: Day 14
Population: All patients that completed the required days of dosing to study end
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 10 mg | 50 mg | 250 mg | 500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5
h*ng/mL | 423 (17.1) | 2240 (23.4) | 14500 (17.9) | 36000 (41.7)

4. Primary Outcome: Pharmacokinetics: Day 1 Plasma Cmax Values
Description: All subjects who completed sample collections for Day 1 plasma N91115
Time Frame: Day 1
Population: All subjects that completed the plasma collection sampling were included in the analysis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 10 mg | 50 mg | 250 mg | 500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5
ng/mL | 33.0 (32.2) | 245 (55.4) | 1810 (50.2) | 3840 (39.6)

5. Primary Outcome: Pharmacokinetics: Plasma Cmax Values on Day 14
Description: Plasma Cmax values from Day 14 subjects with repeat administration of N91115
Time Frame: Day 14
Population: All subjects completing plasma collection sampling for N91115
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 10 mg | 50 mg | 250 mg | 500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5
ng/mL | 84.3 (44.4) | 445 (48.6) | 2410 (30.3) | 5800 (67.2)

ADVERSE EVENTS:
Time Frame: AEs were collected from the time of informed consent for the study duration (up to 14 days) and during a non-dosing period of 7 days afterwards.
Description: Treatment emergent adverse event (TEAE), defined as AEs that are not present prior to the start of study medication, or present before study medication that worsened after starting study medication. TEAEs may be related to study or a procedure conducted during the study.
  Subject is counted only once within System organ class and preferred term.
Arm/Group | Placebo | 10 mg | 50 mg | 250 mg | 500 mg | 50 mg (Single Dose) | 250 mg (Fed) | Placebo- Single Dose
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 9/9 | 6/6 | 6/6 | 6/6 | 6/6 | 1/6 | 4/6 | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=9) | 10 mg (N=6) | 50 mg (N=6) | 250 mg (N=6) | 500 mg (N=6) | 50 mg (Single Dose) (N=6) | 250 mg (Fed) (N=6) | Placebo- Single Dose (N=4)
Palpitation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye Pruritus (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous Stomatitis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Change Of Bowel Habit (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft Tissue Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine Odor Abnormal (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 9 (9) | 6 (6) | 6 (6) | 6 (6) | 6 (6) | 0 (0) | 4 (4) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less